CLINICAL TRIAL: NCT02912715
Title: Prospective, Multi-center, Non-randomized Clinical Trial of Passeo-18 Lux Drug Coated Balloon（DCB） in New and Non-stented Re-stenotic Lesions in the Superficial Femoral Artery (SFA) and Proximal Popliteal Artery (PPA) in a Chinese Patient Population
Brief Title: BIOLUX P-IV CHINA ( BIOTRONIK )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik (Beijing) Medical Device Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1303
Record Dates: First submitted 2016-09-08; First posted 2016-09-23 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2022-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel releasing angioplasty balloon (Experimental): Intervention treatment of balloon angioplasty with Paclitaxel releasing angioplasty balloon(Passeo-18 Lux) in new and non-stented re-stenotic lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA)
  Interventions: Device: Paclitaxel releasing angioplasty balloon

INTERVENTIONS:
Device: Paclitaxel releasing angioplasty balloon — Paclitaxel releasing angioplasty balloon catheter is advanced through an introducer sheath and tracked over the wire until reaching the target lesion. The balloon can be precisely positioned by means of the radiopaque markers crimped on the inner shaft of the catheter. The catheter is dilated up to its intended diameter by inflating the balloon with a solution containing contrast media, causing a compression of the arterial plaque against the inner lining of the arterial wall and improving blood flow. After balloon inflation, the drug-carrier adheres to the arterial wall and facilitates the drug release to surrounding tissue. As there is no need for sustained release of Paclitaxel after the inflation, the drug carrier dissolves rapidly.

SUMMARY:
Prospective, multi-center, non-randomized clinical trial with follow-up investigations at 1, 6 and 12 months. To confirm safety and efficacy of Passeo-18 Lux DCB in new and non-stented re-stenotic lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) in a Chinese patient population.

DETAILED DESCRIPTION:
A prospective, multi-centre, non-randomized clinical trial with follow-up investigations at 1, 6 and 12 months. Approximately 158 subjects will be enrolled at 15 Chinese study sites. To confirm the safety and efficacy of the Passeo-18 Lux DCB for the interventional treatment of new and non-stented re-stenotic lesions in the superficial femoral artery (SFA) and proximal popliteal artery (PPA) in a Chinese patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Subject with documented diagnosis of peripheral arterial disease (PAD) classified as Rutherford class 2-3-4 in the superficial femoral artery (SFA) and/or proximal popliteal artery (PPA) above the knee, located in the arterial segment starting at least 1 cm beyond the common femoral artery (CFA) bifurcation between the superficial and profunda femoris arteries (proximal anatomical landmark) to the distal P1 segment of the popliteal artery at the level of the proximal edge of the patella (distal anatomical landmark).
* Subject able to walk without assistive devices (e.g. walker, cane).
* Female subjects of childbearing potential must have a negative pregnancy test ≤ 7 days before index procedure; Both male and female subjects are willing to use a reliable method of birth control for the duration of the study or must have documented adequate birth control.
* Signed and dated Patient Informed Consent (PIC) form.
* Subject understands and accepts the duration of the study and is able and willing to comply with all requirements, including follow-up visits and evaluations.
* Life expectancy, in the Investigator's opinion, of at least 12 months.
* Target lesion consists of a de novo or non-stented restenotic lesion with a ≥70% diameter stenosis.
* Lesion length≤ 200 mm.
* Reference vessel diameter ≥ 2 mm and ≤ 7 mm by visual estimate.
* Subject with ipsilateral/contralateral iliac disease that requires treatment during the index procedure can be included if treatment is successful (angiographic evidence of stenosis <30%). Iliac disease should be treated firstly by marketed devices excluding drug eluted stent and drug coated balloon.
* Angiographic evidence of adequate distal run-off to the foot (at least one native calf vessel [posterior tibial, anterior tibial, or peroneal arteries] is patent, defined as < 50% diameter stenosis).

Exclusion Criteria:

* Stroke or STEMI within 3 months prior to index procedure.
* Either local or systemic thrombolytic therapy within 48 hours prior to index procedure.
* Inability to tolerate oral anticoagulation therapy (blood thinners such as warfarin) while on concomitant dual antiplatelet therapy (DAPT).
* Known allergies or sensitivities to heparin, aspirin (ASA), other anticoagulant/anti-platelet therapies, and/or paclitaxel or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
* Breastfeeding women.
* Chronic renal insufficiency with serum creatinine > 2.5 mg/dL within 14 days prior to index procedure.
* White blood cell count (WBC) < 3,000 cells/mm3 within 14 days prior to index procedure.
* Platelet count < 80,000 cells/mm3 or > 700,000 cells/mm3 within 14 days prior to index procedure.
* Known or suspected active systemic infection evidenced by WBC > 14.0 (14000/mm3) within 14 days prior to index procedure.
* Diagnosed with bleeding diatheses or hypercoagulable state.
* Subject is enrolled in any investigational device, drug or biologic study.
* Any major (e.g., cardiac. peripheral, abdominal) surgical procedure or planned intervention performed within 30 days prior to the index procedure.
* Any major (e.g., cardiac. peripheral, abdominal) elective procedure or intervention within 30 days post index procedure.
* Target lesion known in advance of enrollment to require treatment with alternative therapy such as (drug-eluting) stent, laser, atherectomy, cryoplasty, re-entry devices, cutting/scoring balloon, brachytherapy. Use of embolic protection devices is also prohibited.
* Contralateral SFA/PPA disease requiring treatment in the same setting as index procedure.
* Presence of additional lesions in the target vessel that require treatment during index procedure but do not meet the inclusion criteria.
* Complete occlusion lesion> 100mm.
* Target lesion is an in-stent or post-DCB restenosis or has been previously treated with bypass surgery.
* Lesion within or adjacent to an aneurysm.
* Acute or sub-acute thrombus in the target vessel.
* Angiographic evidence of severe calcification.
* Failure to successfully cross the target lesion with a guide wire.
* Pre-dilation resulted in a major (≥ Grade D) flow-limiting dissection (observed on 2 orthogonal views) or residual stenosis > 70% or translesional peak gradient > 10mm Hg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 12 months
  a composite of device- and procedure-related mortality, major target limb amputation and clinically-driven target lesion revascularization（TLR） within 12-months post-initial procedure.

SECONDARY OUTCOMES:
Death of any cause | 30 days, 6 and 12 months
  the all-cause mortality of subjects at 30 days, 6 months and 12 months after index procedure
Target lesion revascularization | 30 days, 6 and 12 months
  TLR,Target lesion revascularization.In the subjects experiencing target lesion revascularization, the two revascularizations were both judged as clinically driven target lesion revascularization.
Clinically-driven target lesion revascularization | 30 days, 6 and 12 months
  Defined as any re-intervention at the target lesion due to symptoms or drop of ABI/TBI of≥20% or >0.15 when compared to post-procedure baseline ABI/TBI（Ankle Brachial Index/Toe Brachial Index）. Clinically driven TLR will be adjudicated by an independent Clinical Event Committee
Target vessel revascularization | 30 days, 6 and 12 months
  TVR,Target vessel revascularization.The target vessel revascularization of subjects at 30 days, 6 months, and 12 months after index procedure.Defined as any re-intervention at the target vessel due to symptoms or drop of ABI/TBI of≥20% or >0.15 when compared to post-procedure baseline ABI/TBI. Clinically driven TVR will be adjudicated by an independent Clinical Event Committee
Clinically-driven target vessel revascularization | 30 days, 6 and 12 months
  Defined as any re-intervention at the target vessel due to symptoms or drop of ABI/TBI of≥20% or >0.15 when compared to post-procedure baseline ABI/TBI. Clinically driven TVR will be adjudicated by an independent Clinical Event Committee
Major target limb amputation | 30 days, 6 and 12 months
  Surgical removal of tissue within the affected limb.
  * Above-knee amputation: amputation at a point above the knee
  * Below-knee amputation: amputation at a point below the knee
Thrombosis at the target lesion site | 30 days, 6 and 12 months
  Rapidly developing into total occlusion due to thrombosis confirmed by sudden onset of symptoms and recorded by Doppler ultrasound and/or angiography. Thrombosis can be classified as acute (<1 day), subacute (1-30 days) and late (> 30 days).
Primary sustained clinical improvement | 6 and 12 months
  Primary sustained clinical improvement at 6 months and 12 months after index procedure is defined as sustained upward shift of at least 1 category on Rutherford classification as compared to baseline without further endovascular or surgical revascularization procedure(s) at target lesion.
Secondary sustained clinical improvement | 6 and 12 months
  Secondary sustained clinical improvement at 6 months and 12 months after surgery defined as sustained upward shift of at least 1 category on Rutherford classification as compared to baseline including further endovascular or surgical revascularization procedures at target lesion.
Duplex-defined binary restenosis (PSVR > 2.4) of the target lesion | 6 and 12 months
  Binary restenosis of the target lesion determined by Duplex ultrasound at the time of re-intervention before 6 months and 12 months after index procedure or any prescheduled time point was judged by PSVR > 2.4.
Walking capacity assessment by Walking Impairment Questionnaire | at baseline, 30 days, 6 and 12 months
  Changes in walking ability assessed with the Walking Impairment Questionnaire (WIQ) at baseline, 30 days, 6 months, and 12 months after index procedure.
Walking distance as assessed by 6 Minute Walk Test | at baseline, 30 days, 6 and 12 months
  Changes in the walking distance assessed with the 6-minute walking test (6MWT) at baseline, 30 days, 6 months, and 12 months after index procedure.
Quality of life assessment by EuroQol Five Dimensions（EQ5D） questionnaire | at baseline, 30 days, 6 and 12 months
  Changes in quality of life assessed with the EQ5D questionnaire at baseline, 30 days, 6 months, and 12 months after index procedure.
Device success | during the procedure
  Device success referred to the intact investigational device successfully performing delivery, balloon inflation, deflation, and withdrawal without bursting below the rated burst pressure (RBP).
Procedural success | during the procedure
  Procedural success referred to residual stenosis ≤ 50% (for subjects without stent) or ≤ 30% (for subjects with stent) as accessed by the core laboratory.
Clinical success | during the hospitalization
  Clinical success, defined as procedural success without procedural complications (death, major target limb amputation, thrombosis of the target lesion, or TVR) prior to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Fu, Principal Investigator — Fudan University
Locations (1):
- Fudan University affiliated Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Derived] Yang J, Yue J, Chen X, Wang H, Jiang W, Huang X, Lu X, Dong H, Li X, Fu W. Safety and Efficacy of the Passeo-18 Lux Drug-Coated Balloon Catheter in Atherosclerotic Femoropopliteal Lesions: The Multicenter BIOLUX P-IV China Study. Ann Vasc Surg. 2023 Jul;93:275-282. doi: 10.1016/j.avsg.2023.01.040. Epub 2023 Feb 14. PMID 36796585
- See also: test link — http://www.ncbi.nlm.nih.gov/pubmed/